CLINICAL TRIAL: NCT05870111
Title: Neurobehavioral and Immune Effects of Citicoline in Youth Alcohol Use Disorder
Brief Title: Citicoline in Youth Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Lindsay Squeglia, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00128800
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder
Keywords: Citicoline
MeSH Terms: conditions — Alcoholism | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citicoline (Experimental): 2000mg/day citicoline for 4 weeks, administered orally
  Interventions: Drug: Citicoline (cytidine diphosphate-choline)
- Placebo (Placebo Comparator): placebo capsule daily for 4 weeks, matched in appearance to citicoline to preserve double-blind, administered orally
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Citicoline (cytidine diphosphate-choline) — 2000mg/day citicoline, administered orally, for 4 weeks
  Arms: Citicoline
Drug: Placebo oral capsule — placebo capsule daily for 4 weeks, matched in appearance to citicoline to preserve double-blind, administered orally
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate how citicoline, an over-the-counter supplement, versus a placebo pill (i.e., an inactive pill) affects the immune system, brain, and cognition in adolescents who may use alcohol.

ELIGIBILITY:
Inclusion:

Age 16 to 22.

Call study team for additional screening and information.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Peripheral Cytokine: IL-1B | 4 weeks of treatment
  Peripheral cytokine (IL-1B) to measure neuroinflammation.
Peripheral Cytokine: IL-6 | 4 weeks of treatment
  Peripheral cytokine (IL-6) to measure neuroinflammation.
Peripheral Cytokine: TNFα | 4 weeks of treatment
  Peripheral cytokine (TNFα) to measure neuroinflammation.
Brain Metabolite: N-acetyl-aspartate | 4 weeks of treatment
  Magnetic resonance spectroscopy to quantify neurometabolites (N-acetyl-aspartate) in the anterior cingulate.
Brain Metabolite: Choline | 4 weeks of treatment
  Magnetic resonance spectroscopy to quantify neurometabolites (choline) in the anterior cingulate.
Neurocognition: Behavioral impulsivity | 4 weeks of treatment
  Behavioral impulsivity will be measured via the Behavioral Approach/Avoidance Scales (BIS/BAS).
Neurocognition: Cognitive Flexibility and Attention | 4 weeks of treatment
  Cognitive flexibility and attention will be measured via the NIH Toolbox Dimensional Change Card Sort.
Neurocognition: Inhibitory Control and Attention | 4 weeks of treatment
  Inhibitory control and attention will be measured via the NIH Toolbox Flanker Inhibitory Control and Attention.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No